CLINICAL TRIAL: NCT03136497
Title: Phase Ib Dose Finding Study of ABT-199 (A-1195425.0) Plus Ibrutinib (PCI-32765) and Rituximab in Patients With Relapsed/Refractory Diffuse Large B-cell NHL (DLBCL)
Brief Title: A Study of ABT-199 Plus Ibrutinib and Rituximab in Patients With Relapsed/Refractory Diffuse Large B-cell Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Hackensack Meridian Health (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00005671; 54179060LYM1004 (Other: Janssen Scientific Affairs, LLC); ML30063 (Other: Genentech, Inc.)
Record Dates: First submitted 2017-04-20; First posted 2017-05-02 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-06

CONDITIONS: Relapsed Diffuse Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — venetoclax; ibrutinib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 400mg ABT-199 (Experimental): Cycle length will be 28 days. 400mg ABT-199 will be administered orally QD (Once Daily), continuously for 24 cycles. Ibrutinib will be administered orally QD, continuously for 24 cycles. Rituximab will be administered IV per institutional standards. weekly X 4 (Cycle 1); once on Day 1 of cycles 2-6 only, then every other cycle until Cycle 24 (total 18 doses of Rituxan from C1D1), Commercially available rituximab IV will be used.
  Interventions: Drug: 400mg ABT-199; Drug: Ibrutinib; Drug: Rituximab
- 800mg ABT-199 (Experimental): Cycle length will be 28 days. 800mg ABT-199 will be administered orally QD (Once Daily), continuously for 24 cycles. Ibrutinib will be administered orally QD, continuously for 24 cycles. Rituximab will be administered IV per institutional standards. weekly X 4 (Cycle 1); once on Day 1 of cycles 2-6 only, then every other cycle until Cycle 24 (total 18 doses of Rituxan from C1D1), Commercially available rituximab IV will be used.
  Interventions: Drug: Ibrutinib; Drug: Rituximab; Drug: 800mg ABT-199

INTERVENTIONS:
Drug: 400mg ABT-199 — Oral dose daily until disease progression
  Other Names: A-1195425.0; Venetoclax
  Arms: 400mg ABT-199
Drug: Ibrutinib — Oral dose daily until disease progression
  Other Names: PIC-32765; Imbruvica
Drug: Rituximab — Rituximab will be administered IV per institutional standards. weekly X 4 (Cycle 1); once on Day 1 of cycles 2-6 only, then every other cycle until Cycle 24 (total 18 doses of Rituxan from C1D1
  Other Names: Rituxan
Drug: 800mg ABT-199 — Oral dose daily until disease progression
  Other Names: A-1195425.0; Venetoclax
  Arms: 800mg ABT-199

SUMMARY:
A Study of Venetoclax Plus Ibrutinib and Rituximab in Patients with Relapsed/Refractory Diffuse Large B-cell Lymphoma (DLBCL).

Our hypothesis is that the combination therapy of BTK (Bruton's tyrosine kinase) Inhibitor Ibrutinib plus Venetoclax and Rituximab in relapsed or refractory DLBCL will have an increased activity with acceptable toxicity. Furthermore, this new novel therapeutic combination will be safe and well tolerated among this patient population.

DETAILED DESCRIPTION:
This is a Phase 1b, single-arm, open-label, single-center study of venetoclax (ABT-199) in combination with ibrutinib and rituximab in Subjects with Relapsed/Refractory DLBCL. The trial consists of a dose-escalation of venetoclax in combination with standard doses of ibrutinib and rituximab. For the dose escalation part of the study, a standard 3+3 design will be utilized. Once the MTD has been established, the dose escalation part will be followed by a dose expansion part in a cohort with a maximum of 24 subjects with DLBCL. The purpose of the dose expansion part is to investigate the efficacy of the combination. Between the dose-escalation and dose-expansion, the maximum number of subjects will be 30.

Cycle length will be 28 days. Venetoclax will be administered orally QD (Once Daily), continuously for 24 cycles. Ibrutinib will be administered orally QD, continuously for 24 cycles. Rituximab will be administered IV per institutional standards. weekly X 4 (Cycle 1); once on Day 1 of cycles 2-6 only, then every other cycle until Cycle 24 (total 18 doses of Rituxan from C1D1), Commercially available rituximab IV will be used.

ELIGIBILITY:
Inclusion Criteria:

* ECOG (Eastern Cooperative Oncology Group) Performance Status </= 2.
* Histologically or cytologically confirmed diagnosis of advanced DLBCL.
* Ability and willingness to comply with the requirements of the study protocol
* Prior therapy: relapsed or refractory patients who have received one prior therapy are eligible. If treated with small molecule, washout therapy with a period of greater than 5 times the half-life of the molecule. Patients who have previously received high-dose chemotherapy with peripheral stem cell support are eligible. Washout period of 21 days.
* Presence of at least one lymph node evaluable or mass measurable for response.
* Age greater than or equal to 18 years.
* Recovery from any previous treatment therapy.
* Laboratory parameters:
* Absolute neutrophil count (ANC) 1000/mm3 independent of growth factor support (unless the treating physician deems the neutropenia is related to bone marrow involvement, then an ANC of > 750/mm3 is allowed)
* Platelets 100,000/mm3 or 50,000/mm3 if bone marrow involvement independent of transfusion support in either situation
* Total bilirubin ≤ 1.5 x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin
* Aspartate Aminotransferase (AST, SGOT) and Alanine Aminotransferase (ALT, SGPT) ≤ 3 x upper limit of normal (ULN)
* Creatinine: Creatinine Clearance (CrCl) 50 ml/min (calculated using Cockcroft-Gault Formula-Appendix 2) -Prothrombin time (PT)or international normalized ratio and partial thromboplastin time (PTT) not to exceed 1.2 times the institution's normal range
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. For females, these restrictions apply for 3 months after Venetoclax and 12 months after Rituximab For males, these restrictions apply for 3 months after the last dose of study drug.
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [-hCG]) or urine pregnancy test at Screening. Women who are pregnant or breastfeeding are ineligible for this study.
* Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study

Exclusion Criteria:

* Known central nervous system lymphoma.
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon).
* Received the following agents within 7 days prior to the first dose of venetoclax or requires chronic treatment with strong Cytochrome P450 3A4 (CYP3A) inhibitors (e.g., ketoconazole, ritonavir, clarithromycin, itraconazole, voriconazole), moderate CYP3A inhibitors (e.g., erythromycin, ciprofloxacin, diltiazem, fluconazole, verapamil), strong CYP3A inducers (e.g., carbamazepine, phenytoin, rifampin, St. John's wort) or moderate CYP3A inducers (e.g., bosentan, efavirenz, etravirine). (See Appendix 4)
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
* Vaccinated with live, attenuated vaccines within 4 weeks of randomization.
* Use of any other standard chemotherapy, radiation therapy, or experimental drug therapy for the treatment of DLBCL within 21 days of starting treatment
* Known history of human immunodeficiency virus (HIV) or active Hepatitis C Virus or active Hepatitis B Virus infection or any uncontrolled active systemic infection or human T-cell leukemia virus 1 (HTLV-1) seropositive status
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, venetoclax or rituximab or put the study outcomes at undue risk.
* History of uncontrolled or symptomatic angina
* Ejection fraction below the institutional normal limit
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* Patients with a history of curatively treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix are generally eligible. Patients with a malignancy that has been treated, but not with curative intent, will also be excluded, unless the malignancy has been in remission without treatment for 2 years prior to enrollment.
* Evidence of other clinically significant uncontrolled condition(s) including, but not limited to, uncontrolled systemic infection (viral, bacterial, or fungal)
* Major surgery (within 4 weeks prior to the start of the first dose of study treatment), other than for diagnosis
* Women who are pregnant or lactating
* Female patients who are not surgically sterile or postmenopausal (for at least 1 year) must practice at least one of the following methods of birth control throughout the duration of study participation and for at least 12 months after study treatment:
* Total abstinence from sexual intercourse
* A vasectomized partner
* Hormonal contraceptives (oral, parenteral, vaginal ring, or transdermal) that started at least 3 months prior to study drug administration
* Double-barrier method (condom diaphragm or cervical cup with spermicidal contraceptive sponge, jellies, or cream)
* Non-vasectomized male patients must comply with at least one of the following methods of birth control throughout the duration of study participation and for at least 12 months after study treatment:
* A partner who is surgically sterile or postmenopausal (for at least 1 year) or who is taking hormonal contraceptives (oral, parenteral, vaginal ring, or transdermal) for at least 3 months prior to study drug administration
* Total abstinence from sexual intercourse
* Double-barrier method (condom diaphragm or cervical cup with spermicidal, contraceptive sponge, jellies, or cream)
* Malabsorption syndrome or other condition that precludes enteral route of administration
* Known allergy to both xanthine oxidase inhibitors and rasburicase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre Goy, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borner C. The Bcl-2 protein family: sensors and checkpoints for life-or-death decisions. Mol Immunol. 2003 Jan;39(11):615-47. doi: 10.1016/s0161-5890(02)00252-3. PMID 12493639
- [Background] Binet JL, Auquier A, Dighiero G, Chastang C, Piguet H, Goasguen J, Vaugier G, Potron G, Colona P, Oberling F, Thomas M, Tchernia G, Jacquillat C, Boivin P, Lesty C, Duault MT, Monconduit M, Belabbes S, Gremy F. A new prognostic classification of chronic lymphocytic leukemia derived from a multivariate survival analysis. Cancer. 1981 Jul 1;48(1):198-206. doi: 10.1002/1097-0142(19810701)48:13.0.co;2-v. PMID 7237385
- [Background] Cairo MS, Bishop M. Tumour lysis syndrome: new therapeutic strategies and classification. Br J Haematol. 2004 Oct;127(1):3-11. doi: 10.1111/j.1365-2141.2004.05094.x. PMID 15384972
- [Background] Calin GA, Cimmino A, Fabbri M, Ferracin M, Wojcik SE, Shimizu M, Taccioli C, Zanesi N, Garzon R, Aqeilan RI, Alder H, Volinia S, Rassenti L, Liu X, Liu CG, Kipps TJ, Negrini M, Croce CM. MiR-15a and miR-16-1 cluster functions in human leukemia. Proc Natl Acad Sci U S A. 2008 Apr 1;105(13):5166-71. doi: 10.1073/pnas.0800121105. Epub 2008 Mar 24. PMID 18362358
- [Background] Catovsky D, Richards S, Matutes E, Oscier D, Dyer M, Bezares RF, Pettitt AR, Hamblin T, Milligan DW, Child JA, Hamilton MS, Dearden CE, Smith AG, Bosanquet AG, Davis Z, Brito-Babapulle V, Else M, Wade R, Hillmen P; UK National Cancer Research Institute (NCRI) Haematological Oncology Clinical Studies Group; NCRI Chronic Lymphocytic Leukaemia Working Group. Assessment of fludarabine plus cyclophosphamide for patients with chronic lymphocytic leukaemia (the LRF CLL4 Trial): a randomised controlled trial. Lancet. 2007 Jul 21;370(9583):230-239. doi: 10.1016/S0140-6736(07)61125-8. PMID 17658394
- [Background] Cheson BD, Bennett JM, Grever M, Kay N, Keating MJ, O'Brien S, Rai KR. National Cancer Institute-sponsored Working Group guidelines for chronic lymphocytic leukemia: revised guidelines for diagnosis and treatment. Blood. 1996 Jun 15;87(12):4990-7. No abstract available. PMID 8652811
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753
- [Background] Coiffier B, Lepage E, Briere J, Herbrecht R, Tilly H, Bouabdallah R, Morel P, Van Den Neste E, Salles G, Gaulard P, Reyes F, Lederlin P, Gisselbrecht C. CHOP chemotherapy plus rituximab compared with CHOP alone in elderly patients with diffuse large-B-cell lymphoma. N Engl J Med. 2002 Jan 24;346(4):235-42. doi: 10.1056/NEJMoa011795. PMID 11807147
- [Background] Coiffier B, Thieblemont C, Van Den Neste E, Lepeu G, Plantier I, Castaigne S, Lefort S, Marit G, Macro M, Sebban C, Belhadj K, Bordessoule D, Ferme C, Tilly H. Long-term outcome of patients in the LNH-98.5 trial, the first randomized study comparing rituximab-CHOP to standard CHOP chemotherapy in DLBCL patients: a study by the Groupe d'Etudes des Lymphomes de l'Adulte. Blood. 2010 Sep 23;116(12):2040-5. doi: 10.1182/blood-2010-03-276246. Epub 2010 Jun 14. PMID 20548096
- [Background] Cory S, Adams JM. The Bcl2 family: regulators of the cellular life-or-death switch. Nat Rev Cancer. 2002 Sep;2(9):647-56. doi: 10.1038/nrc883. PMID 12209154
- [Background] Cory S, Huang DC, Adams JM. The Bcl-2 family: roles in cell survival and oncogenesis. Oncogene. 2003 Nov 24;22(53):8590-607. doi: 10.1038/sj.onc.1207102. PMID 14634621
- [Background] Davis RE, Ngo VN, Lenz G, Tolar P, Young RM, Romesser PB, Kohlhammer H, Lamy L, Zhao H, Yang Y, Xu W, Shaffer AL, Wright G, Xiao W, Powell J, Jiang JK, Thomas CJ, Rosenwald A, Ott G, Muller-Hermelink HK, Gascoyne RD, Connors JM, Johnson NA, Rimsza LM, Campo E, Jaffe ES, Wilson WH, Delabie J, Smeland EB, Fisher RI, Braziel RM, Tubbs RR, Cook JR, Weisenburger DD, Chan WC, Pierce SK, Staudt LM. Chronic active B-cell-receptor signalling in diffuse large B-cell lymphoma. Nature. 2010 Jan 7;463(7277):88-92. doi: 10.1038/nature08638. PMID 20054396
- [Background] Del Gaizo Moore V, Brown JR, Certo M, Love TM, Novina CD, Letai A. Chronic lymphocytic leukemia requires BCL2 to sequester prodeath BIM, explaining sensitivity to BCL2 antagonist ABT-737. J Clin Invest. 2007 Jan;117(1):112-21. doi: 10.1172/JCI28281. PMID 17200714
- [Background] Del Gaizo Moore V, Letai A. Rational design of therapeutics targeting the BCL-2 family: are some cancer cells primed for death but waiting for a final push? Adv Exp Med Biol. 2008;615:159-75. doi: 10.1007/978-1-4020-6554-5_8. PMID 18437895
- [Background] Dighiero G, Binet JL. When and how to treat chronic lymphocytic leukemia. N Engl J Med. 2000 Dec 14;343(24):1799-801. doi: 10.1056/NEJM200012143432410. No abstract available. PMID 11114321
- [Background] Eichhorst BF, Busch R, Hopfinger G, Pasold R, Hensel M, Steinbrecher C, Siehl S, Jager U, Bergmann M, Stilgenbauer S, Schweighofer C, Wendtner CM, Dohner H, Brittinger G, Emmerich B, Hallek M; German CLL Study Group. Fludarabine plus cyclophosphamide versus fludarabine alone in first-line therapy of younger patients with chronic lymphocytic leukemia. Blood. 2006 Feb 1;107(3):885-91. doi: 10.1182/blood-2005-06-2395. Epub 2005 Oct 11. PMID 16219797
- [Background] Feugier P, Van Hoof A, Sebban C, Solal-Celigny P, Bouabdallah R, Ferme C, Christian B, Lepage E, Tilly H, Morschhauser F, Gaulard P, Salles G, Bosly A, Gisselbrecht C, Reyes F, Coiffier B. Long-term results of the R-CHOP study in the treatment of elderly patients with diffuse large B-cell lymphoma: a study by the Groupe d'Etude des Lymphomes de l'Adulte. J Clin Oncol. 2005 Jun 20;23(18):4117-26. doi: 10.1200/JCO.2005.09.131. Epub 2005 May 2. PMID 15867204
- [Background] Flinn IW, Neuberg DS, Grever MR, Dewald GW, Bennett JM, Paietta EM, Hussein MA, Appelbaum FR, Larson RA, Moore DF Jr, Tallman MS. Phase III trial of fludarabine plus cyclophosphamide compared with fludarabine for patients with previously untreated chronic lymphocytic leukemia: US Intergroup Trial E2997. J Clin Oncol. 2007 Mar 1;25(7):793-8. doi: 10.1200/JCO.2006.08.0762. Epub 2007 Feb 5. PMID 17283364
- [Background] Mathews Griner LA, Guha R, Shinn P, Young RM, Keller JM, Liu D, Goldlust IS, Yasgar A, McKnight C, Boxer MB, Duveau DY, Jiang JK, Michael S, Mierzwa T, Huang W, Walsh MJ, Mott BT, Patel P, Leister W, Maloney DJ, Leclair CA, Rai G, Jadhav A, Peyser BD, Austin CP, Martin SE, Simeonov A, Ferrer M, Staudt LM, Thomas CJ. High-throughput combinatorial screening identifies drugs that cooperate with ibrutinib to kill activated B-cell-like diffuse large B-cell lymphoma cells. Proc Natl Acad Sci U S A. 2014 Feb 11;111(6):2349-54. doi: 10.1073/pnas.1311846111. Epub 2014 Jan 27. PMID 24469833
- [Background] Hallek M, Cheson BD, Catovsky D, Caligaris-Cappio F, Dighiero G, Dohner H, Hillmen P, Keating MJ, Montserrat E, Rai KR, Kipps TJ; International Workshop on Chronic Lymphocytic Leukemia. Guidelines for the diagnosis and treatment of chronic lymphocytic leukemia: a report from the International Workshop on Chronic Lymphocytic Leukemia updating the National Cancer Institute-Working Group 1996 guidelines. Blood. 2008 Jun 15;111(12):5446-56. doi: 10.1182/blood-2007-06-093906. Epub 2008 Jan 23. PMID 18216293
- [Background] Habermann TM, Weller EA, Morrison VA, Gascoyne RD, Cassileth PA, Cohn JB, Dakhil SR, Woda B, Fisher RI, Peterson BA, Horning SJ. Rituximab-CHOP versus CHOP alone or with maintenance rituximab in older patients with diffuse large B-cell lymphoma. J Clin Oncol. 2006 Jul 1;24(19):3121-7. doi: 10.1200/JCO.2005.05.1003. Epub 2006 Jun 5. PMID 16754935
- [Background] Hillmen P, Skotnicki AB, Robak T, Jaksic B, Dmoszynska A, Wu J, Sirard C, Mayer J. Alemtuzumab compared with chlorambucil as first-line therapy for chronic lymphocytic leukemia. J Clin Oncol. 2007 Dec 10;25(35):5616-23. doi: 10.1200/JCO.2007.12.9098. Epub 2007 Nov 5. PMID 17984186
- [Background] Howard SC, Jones DP, Pui CH. The tumor lysis syndrome. N Engl J Med. 2011 May 12;364(19):1844-54. doi: 10.1056/NEJMra0904569. No abstract available. PMID 21561350
- [Background] Johnson S, Smith AG, Loffler H, Osby E, Juliusson G, Emmerich B, Wyld PJ, Hiddemann W. Multicentre prospective randomised trial of fludarabine versus cyclophosphamide, doxorubicin, and prednisone (CAP) for treatment of advanced-stage chronic lymphocytic leukaemia. The French Cooperative Group on CLL. Lancet. 1996 May 25;347(9013):1432-8. doi: 10.1016/s0140-6736(96)91681-5. PMID 8676625
- [Background] Korsmeyer SJ. BCL-2 gene family and the regulation of programmed cell death. Cancer Res. 1999 Apr 1;59(7 Suppl):1693s-1700s. PMID 10197582
- [Background] Leporrier M, Chevret S, Cazin B, Boudjerra N, Feugier P, Desablens B, Rapp MJ, Jaubert J, Autrand C, Divine M, Dreyfus B, Maloum K, Travade P, Dighiero G, Binet JL, Chastang C; French Cooperative Group on Chronic Lymphocytic Leukemia. Randomized comparison of fludarabine, CAP, and ChOP in 938 previously untreated stage B and C chronic lymphocytic leukemia patients. Blood. 2001 Oct 15;98(8):2319-25. doi: 10.1182/blood.v98.8.2319. PMID 11588025
- [Background] Matutes E, Polliack A. Morphological and immunophenotypic features of chronic lymphocytic leukemia. Rev Clin Exp Hematol. 2000 Mar;4(1):22-47. doi: 10.1046/j.1468-0734.2000.00002.x. PMID 11486329
- [Background] Moller MB, Pedersen NT, Christensen BE. Mantle cell lymphoma: prognostic capacity of the Follicular Lymphoma International Prognostic Index. Br J Haematol. 2006 Apr;133(1):43-9. doi: 10.1111/j.1365-2141.2006.05970.x. PMID 16512827
- [Background] Oldereid NB, Angelis PD, Wiger R, Clausen OP. Expression of Bcl-2 family proteins and spontaneous apoptosis in normal human testis. Mol Hum Reprod. 2001 May;7(5):403-8. doi: 10.1093/molehr/7.5.403. PMID 11331661
- [Background] Pfreundschuh M, Trumper L, Osterborg A, Pettengell R, Trneny M, Imrie K, Ma D, Gill D, Walewski J, Zinzani PL, Stahel R, Kvaloy S, Shpilberg O, Jaeger U, Hansen M, Lehtinen T, Lopez-Guillermo A, Corrado C, Scheliga A, Milpied N, Mendila M, Rashford M, Kuhnt E, Loeffler M; MabThera International Trial Group. CHOP-like chemotherapy plus rituximab versus CHOP-like chemotherapy alone in young patients with good-prognosis diffuse large-B-cell lymphoma: a randomised controlled trial by the MabThera International Trial (MInT) Group. Lancet Oncol. 2006 May;7(5):379-91. doi: 10.1016/S1470-2045(06)70664-7. PMID 16648042
- [Background] Rai KR, Peterson BL, Appelbaum FR, Kolitz J, Elias L, Shepherd L, Hines J, Threatte GA, Larson RA, Cheson BD, Schiffer CA. Fludarabine compared with chlorambucil as primary therapy for chronic lymphocytic leukemia. N Engl J Med. 2000 Dec 14;343(24):1750-7. doi: 10.1056/NEJM200012143432402. PMID 11114313
- [Background] Roberts AW, Seymour JF, Brown JR, Wierda WG, Kipps TJ, Khaw SL, Carney DA, He SZ, Huang DC, Xiong H, Cui Y, Busman TA, McKeegan EM, Krivoshik AP, Enschede SH, Humerickhouse R. Substantial susceptibility of chronic lymphocytic leukemia to BCL2 inhibition: results of a phase I study of navitoclax in patients with relapsed or refractory disease. J Clin Oncol. 2012 Feb 10;30(5):488-96. doi: 10.1200/JCO.2011.34.7898. Epub 2011 Dec 19. PMID 22184378
- [Background] Rosenwald A, Wright G, Chan WC, Connors JM, Campo E, Fisher RI, Gascoyne RD, Muller-Hermelink HK, Smeland EB, Giltnane JM, Hurt EM, Zhao H, Averett L, Yang L, Wilson WH, Jaffe ES, Simon R, Klausner RD, Powell J, Duffey PL, Longo DL, Greiner TC, Weisenburger DD, Sanger WG, Dave BJ, Lynch JC, Vose J, Armitage JO, Montserrat E, Lopez-Guillermo A, Grogan TM, Miller TP, LeBlanc M, Ott G, Kvaloy S, Delabie J, Holte H, Krajci P, Stokke T, Staudt LM; Lymphoma/Leukemia Molecular Profiling Project. The use of molecular profiling to predict survival after chemotherapy for diffuse large-B-cell lymphoma. N Engl J Med. 2002 Jun 20;346(25):1937-47. doi: 10.1056/NEJMoa012914. PMID 12075054
- [Background] Sehn LH, Donaldson J, Chhanabhai M, Fitzgerald C, Gill K, Klasa R, MacPherson N, O'Reilly S, Spinelli JJ, Sutherland J, Wilson KS, Gascoyne RD, Connors JM. Introduction of combined CHOP plus rituximab therapy dramatically improved outcome of diffuse large B-cell lymphoma in British Columbia. J Clin Oncol. 2005 Aug 1;23(22):5027-33. doi: 10.1200/JCO.2005.09.137. Epub 2005 Jun 13. PMID 15955905
- [Background] Shankland KR, Armitage JO, Hancock BW. Non-Hodgkin lymphoma. Lancet. 2012 Sep 1;380(9844):848-57. doi: 10.1016/S0140-6736(12)60605-9. Epub 2012 Jul 25. PMID 22835603
- [Background] Shustik C, Mick R, Silver R, Sawitsky A, Rai K, Shapiro L. Treatment of early chronic lymphocytic leukemia: intermittent chlorambucil versus observation. Hematol Oncol. 1988 Jan-Mar;6(1):7-12. doi: 10.1002/hon.2900060103. PMID 3277904
- [Background] Smith TJ, Khatcheressian J, Lyman GH, Ozer H, Armitage JO, Balducci L, Bennett CL, Cantor SB, Crawford J, Cross SJ, Demetri G, Desch CE, Pizzo PA, Schiffer CA, Schwartzberg L, Somerfield MR, Somlo G, Wade JC, Wade JL, Winn RJ, Wozniak AJ, Wolff AC. 2006 update of recommendations for the use of white blood cell growth factors: an evidence-based clinical practice guideline. J Clin Oncol. 2006 Jul 1;24(19):3187-205. doi: 10.1200/JCO.2006.06.4451. Epub 2006 May 8. PMID 16682719
- [Background] Sugiyama N, Obinata M, Matsui Y. Bcl-2 inhibits apoptosis of spermatogonia and growth of spermatogonial stem cells in a cell-intrinsic manner. Mol Reprod Dev. 2001 Jan;58(1):30-8. doi: 10.1002/1098-2795(200101)58:13.0.CO;2-4. PMID 11144217
- [Background] Thurmes P, Call T, Slager S, Zent C, Jenkins G, Schwager S, Bowen D, Kay N, Shanafelt T. Comorbid conditions and survival in unselected, newly diagnosed patients with chronic lymphocytic leukemia. Leuk Lymphoma. 2008 Jan;49(1):49-56. doi: 10.1080/10428190701724785. PMID 18203011
- [Background] Vose JM, Link BK, Grossbard ML, Czuczman M, Grillo-Lopez A, Gilman P, Lowe A, Kunkel LA, Fisher RI. Phase II study of rituximab in combination with chop chemotherapy in patients with previously untreated, aggressive non-Hodgkin's lymphoma. J Clin Oncol. 2001 Jan 15;19(2):389-97. doi: 10.1200/JCO.2001.19.2.389. PMID 11208830
- [Background] Wang ML, Rule S, Martin P, Goy A, Auer R, Kahl BS, Jurczak W, Advani RH, Romaguera JE, Williams ME, Barrientos JC, Chmielowska E, Radford J, Stilgenbauer S, Dreyling M, Jedrzejczak WW, Johnson P, Spurgeon SE, Li L, Zhang L, Newberry K, Ou Z, Cheng N, Fang B, McGreivy J, Clow F, Buggy JJ, Chang BY, Beaupre DM, Kunkel LA, Blum KA. Targeting BTK with ibrutinib in relapsed or refractory mantle-cell lymphoma. N Engl J Med. 2013 Aug 8;369(6):507-16. doi: 10.1056/NEJMoa1306220. Epub 2013 Jun 19. PMID 23782157
- [Background] Weisenburger DD. Epidemiology of non-Hodgkin's lymphoma: recent findings regarding an emerging epidemic. Ann Oncol. 1994;5 Suppl 1:19-24. doi: 10.1093/annonc/5.suppl_1.s19. PMID 8172811
- [Background] Wilson WH, Young RM, Schmitz R, Yang Y, Pittaluga S, Wright G, Lih CJ, Williams PM, Shaffer AL, Gerecitano J, de Vos S, Goy A, Kenkre VP, Barr PM, Blum KA, Shustov A, Advani R, Fowler NH, Vose JM, Elstrom RL, Habermann TM, Barrientos JC, McGreivy J, Fardis M, Chang BY, Clow F, Munneke B, Moussa D, Beaupre DM, Staudt LM. Targeting B cell receptor signaling with ibrutinib in diffuse large B cell lymphoma. Nat Med. 2015 Aug;21(8):922-6. doi: 10.1038/nm.3884. Epub 2015 Jul 20. PMID 26193343
- [Background] Yan W, Huang JX, Lax AS, Pelliniemi L, Salminen E, Poutanen M, Toppari J. Overexpression of Bcl-W in the testis disrupts spermatogenesis: revelation of a role of BCL-W in male germ cell cycle control. Mol Endocrinol. 2003 Sep;17(9):1868-79. doi: 10.1210/me.2002-0389. Epub 2003 Jun 13. PMID 12808071
- [Background] Yancik R. Cancer burden in the aged: an epidemiologic and demographic overview. Cancer. 1997 Oct 1;80(7):1273-83. PMID 9317180

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 Patients Consented (9 started, 1 screen failure)
Groups:
- 400mg ABT-199: 400mg ABT-199 Dose Level
- 800mg ABT-199: 800mg ABT-199 Dose Level
- Dose-Expansion 800mg ABT-199: 800mg ABT-199 Dose Level Expansion Arm
Period: Overall Study
Arm/Group | 400mg ABT-199 | 800mg ABT-199 | Dose-Expansion 800mg ABT-199
Started | 5 | 3 | 2
Completed | 4 | 3 | 2
Not Completed | 1 | 0 | 0
Not completed — Screen Failure | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 10 patients consented, of which 9 were treated and 1 screen failure
Groups:
- Total: Total of all reporting groups
Arm/Group | 400mg ABT-199 | 800mg ABT-199 | Dose-Expansion 800mg ABT-199 | Total
Number analyzed (Participants) | 5 | 3 | 2 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 0 | 3
  >=65 years | 4 | 1 | 2 | 7
Age, Continuous [Median (Full Range); unit: Years] | 70 [44 to 74] | 53 [35 to 77] | 84 [83 to 85] | 71.5 [35 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 3 | 1 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 3 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 2 | 1 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: Define maximum tolerated dose and /or recommended phase II dose for the combinations of venetoclax (ABT-199, GDC-0199) plus Ibrutinib (PCI-32765) and rituximab in Relapsed or Refractory DLBCL by assessing the incidence of dose limiting toxicities (DLTs).
Time Frame: 29 days
Measure: Number; unit: mg
Groups:
- ABT-199 Plus Ibrutinib and Rituximab: Cycle length will be 28 days. Venetoclax will be administered orally QD (Once Daily), continuously for 24 cycles. Ibrutinib will be administered orally QD, continuously for 24 cycles. Rituximab will be administered IV per institutional standards. weekly X 4 (Cycle 1); once on Day 1 of cycles 2-6 only, then every other cycle until Cycle 24 (total 18 doses of Rituxan from C1D1), Commercially available rituximab IV will be used.
  ABT-199: Oral dose daily until disease progression
  Ibrutinib: Oral dose daily until disease progression
  Rituximab: Rituximab will be administered IV per institutional standards. weekly X 4 (Cycle 1); once on Day 1 of cycles 2-6 only, then every other cycle until Cycle 24 (total 18 doses of Rituxan from C1D1
Arm/Group | ABT-199 Plus Ibrutinib and Rituximab
Number analyzed (Participants) | 9
mg | 800

2. Secondary Outcome: Incidence of Treatment-emergent Adverse Events.
Description: Adverse events will be assessed using the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE), version 4.03.
Time Frame: 36 Months
Population: Number of participants with treatment-emergency adverse events
Measure: Count of Participants; unit: Participants
Arm/Group | 400mg ABT-199 | 800mg ABT-199 | Dose-Expansion 800mg ABT-199
Number analyzed (Participants) | 4 | 3 | 2
Participants | 3 | 2 | 1

3. Secondary Outcome: Efficacy as Assessed by Progression Free Survival (PFS)
Description: The duration of PFS is defined as the time from the beginning of the first cycle of treatment to the date of progressive disease or death from any cause. PFS will be estimated using Kaplan-Meier method.
Time Frame: 36 Months
Population: Median Progression Free Survival
Measure: Median (Full Range); unit: Months
Arm/Group | 400mg ABT-199 | 800mg ABT-199 | Dose-Expansion 800mg ABT-199
Number analyzed (Participants) | 3 | 2 | 2
Months | 2 [1 to 4] | 2 [2 to 2] | 2 [1 to 4]

4. Secondary Outcome: Efficacy as Assessed by Overall Survival (OS)
Description: The duration of OS is defined as the time from the beginning of the first cycle of treatment to the date of death from any cause. OS will be estimated using Kaplan-Meier method.
Time Frame: 36 Months
Population: Median Overall Survival
Measure: Median (Full Range); unit: Months
Arm/Group | 400mg ABT-199 | 800mg ABT-199 | Dose-Expansion 800mg ABT-199
Number analyzed (Participants) | 3 | 3 | 2
Months | 8.6 [2.1 to 32.1] | 3.5 [2.1 to 11.2] | 9.4 [9.4 to 9.4]

ADVERSE EVENTS:
Time Frame: 36 Months
Arm/Group | 400mg ABT-199 | 800mg ABT-199 | Dose-Expansion 800mg ABT-199
All-Cause Mortality (participants affected / at risk) | 3/4 | 2/3 | 1/2
Serious Adverse Events (participants affected / at risk) | 3/4 | 1/3 | 1/2
Other Adverse Events (participants affected / at risk) | 3/4 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 400mg ABT-199 (N=4) | 800mg ABT-199 (N=3) | Dose-Expansion 800mg ABT-199 (N=2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoidal Bleed (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Left Hip Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Syncopal Episode (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 400mg ABT-199 (N=4) | 800mg ABT-199 (N=3) | Dose-Expansion 800mg ABT-199 (N=2)
Alk Phosphatase Elevated (Investigations) | 1 (1) | 0 (0) | 0 (0)
Allergies, seasonal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Elevated AST (Investigations) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric Upset (GERD) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headaches (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
LDH Elevated (Investigations) | 0 (0) | 1 (1) | 0 (0)
Localized edema LLE (General disorders) | 1 (1) | 0 (0) | 0 (0)
Loose Bowels (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal Bleed (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/97/NCT03136497/Prot_SAP_000.pdf